CLINICAL TRIAL: NCT01214317
Title: Study of Combinative Effect of Induction Therapy With Mitoxantrone and Plasmapheresis to Treat Patients With Aggressive Multiple Sclerosis
Brief Title: Study of Induction Therapy With Mitoxantrone and Plasmapheresis to Treat Aggressive Multiple Sclerosis
Acronym: IMPAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Etemadifar, Professor of neurology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 389050
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; mitoxantrone; plasmapheresis; induction therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Plasmapheresis; Mitoxantrone; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mitoxantrone and plasmapheresis (Active Comparator): Monthly Plasmapheresis (plasma exchange machine: Haemonetics, model TCS2, USA) 25 ml/kg for 5 cycles, with replacement of 0.9% saline and 5% human serum albumin followed by monthly IV infusion of 12 mg/m2 mitoxantrone (EBEWE Pharma, Amsterdam, The Netherlands) at the end of each Plasmapheresis course for three successive months. Then, treatment is continued by adding two more 6 mg/m2 doses of mitoxantrone in 3-month intervals.
  Interventions: Procedure: plasmapheresis
- mitoxantrone (No Intervention): Monthly IV infusion of 12 mg/m2 mitoxantrone (EBEWE Pharma, Amsterdam, The Netherlands) for three successive months. Then, treatment is continued by adding two more 6 mg/m2 doses of mitoxantrone in 3-month intervals.

INTERVENTIONS:
Procedure: plasmapheresis — 3 courses of plasmapheresis are performed before mitoxantrone injection in first 3 months to investigate the efficacy of plasmapheresis in comparison with the other arm that are only treated with mitoxantrone
  Other Names: novantrone; plasma exchange
  Arms: mitoxantrone and plasmapheresis

SUMMARY:
The purpose of this study is to compare the effect of combinative induction therapy with mitoxantrone and plasmapheresis versus induction therapy with mitoxantrone alone in cases of aggressive multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Aggressive multiple sclerosis in attack phase
* EDSS: 1-5
* No contraindication for mitoxantrone prescription
* No past history of mitoxantrone injection
* No history of corticosteroid and immunosuppressive therapy in last 3 months

Exclusion Criteria:

* Patient's incompliance
* Severe drug induced side effects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Etemadifar, Principal Investigator — Alzahra Hospital
Locations (1):
- Alahra hospital, Isfahan, Iran

RESULTS

PARTICIPANT FLOW:
Groups:
- Mitoxantrone and Plasmapheresis: Monthly plasmapheresis (plasma exchange machine: Haemonetics, model TCS2, USA) 25 ml/kg for 5 cycles, with replacement of 0.9% saline and 5% human serum albumin followed by monthly IV infusion of 12 mg/m2 mitoxantrone (EBEWE Pharma, Amsterdam, The Netherlands) at the end of each plasmapheresis course for three successive months to investigate the efficacy of plasmapheresis in comparison with the other arm that are only treated with mitoxantrone. Then, treatment is continued by adding two more 6 mg/m2 doses of mitoxantrone in 3-month intervals.
Period: Overall Study
Arm/Group | Mitoxantrone and Plasmapheresis | Mitoxantrone
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitoxantrone and Plasmapheresis | Mitoxantrone | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (11.3) | 29.1 (6.7) | 29.68 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Iran | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Expanded Disability Status Score
Description: The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and defines functional systems as pyramidalm, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral and others.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Time Frame: At the end of month 8 after treatment initiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mitoxantrone and Plasmapheresis | Mitoxantrone
Number analyzed (Participants) | 18 | 22
score on a scale | 2.9 (1.3) | 2.6 (0.9)

2. Primary Outcome: Change From Baseline in Mean Number of MS Plaques Found on Brain MRI
Description: Change From Baseline in Mean Number of MS plaques found on Brain MRI 8 months after treatment initiation
Time Frame: Month 8 after treatment initiation
Measure: Mean (Standard Deviation); unit: Plaques
Arm/Group | Mitoxantrone and Plasmapheresis | Mitoxantrone
Number analyzed (Participants) | 18 | 22
Plaques | 3.5 (0.9) | 7.3 (1.6)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Mitoxantrone and Plasmapheresis | Mitoxantrone
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 6/18 | 7/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitoxantrone and Plasmapheresis (N=18) | Mitoxantrone (N=22)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Transient amenorrhea (Reproductive system and breast disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 0 | 1
Transient rise in liver enzymes (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes